CLINICAL TRIAL: NCT07010185
Title: Effect of Supervised Versus Unsupervised Strength Training on Balance and Functional Performance Among Post Stroke Ambulatory Patients: A Single-Blinded Randomized Controlled Study
Brief Title: Effect of Supervised Versus Unsupervised Strength Training on Balance and Functional Performance Among Post Stroke Ambulatory Patients
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHasan; Majmaah University (Registry Identifier: DSR)
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Cerebro-vascular Accident
Keywords: cerebrovascular accident; Stroke; Post Stroke Ambulatory Patients
MeSH Terms: conditions — Stroke | interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: two-arm randomized control approach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supervised training (Experimental): supervised strength training
  Interventions: Behavioral: home based exercise

INTERVENTIONS:
Behavioral: home based exercise — warm-up Exercises (5 minutes), dynamic Stretching (5 to 10 repetitions), strengthening exercises focused on lower limb muscles, such as bridging, clamshells, and various leg exercises (5-10 repetitions across 2-3 sets, based on patient tolerance)
  Other Names: stretching; warm up

SUMMARY:
Objective:

This single-blinded randomized controlled trial compared the effects of supervised clinic-based versus unsupervised home-based balance and strength training on functional outcomes in ambulatory post-stroke patients.

Methods:

This study implemented a single-blinded; two-arm randomized control approach to evaluate rehabilitation interventions for stroke patients. It was conducted at the Prince Sultan Military Medical City in the Riyadh region, which features a specialized physiotherapy center for neurology patients.

Design: RCT with two parallel arms (N=48; 24/group). Participants: Ambulatory stroke survivors (1-24 months post-stroke) aged 25-65 years.

Interventions:

Supervised group: 45-minute therapist-led sessions (3x/week for 12 weeks), including strength/balance exercises.

Unsupervised group: Identical exercises performed at home with remote guidance (videos, diaries, follow-up calls).

Outcomes: Berg Balance Scale (BBS), Physiological Cost Index (PCI), 6-minute walk test (6MWT), and Short Form-36 (SF-36) at baseline and 12 weeks.

DETAILED DESCRIPTION:
Stroke, often referred to as a cerebrovascular accident, is a significant global health concern and a leading cause of long-term disability, particularly among the elderly. Stroke occurs when there is a sudden disruption of blood flow to the brain, causing the death of cerebral tissue [1]. Globally, stroke affects around 15 million individuals each year, resulting in 5 million deaths and 5 million cases of permanent disability, making it a leading cause of mortality and morbidity (World Health Organization). In Europe alone, there are 41.5 million new stroke cases each year, with only 15% of patients achieving full recovery [2]. In Saudi Arabia it remains a significant health concern with an incidence of 29.8 cases per 100,000 individuals annually [3]. The incidence rates of stroke vary regionally, with 15.1 per 100,000 in Jizan city and up to 29.8 per 100,000 in the Eastern region and urban areas experiencing higher rates than rural ones [4, 5]. Although these rates are lower than rates in many high-income countries, there is a pressing need for a nationwide stroke registry to enhance healthcare services for survivors [3]. Ischemic strokes are the most common subtype, while hemorrhagic strokes, particularly those related to hypertension, also present significant challenges [6]. The risk factors for stroke in the Saudi population include hypertension, diabetes mellitus, hypercholesterolemia, obesity, physical inactivity, heredity, and smoking [7]. These factors contribute significantly to the overall burden of stroke and highlight the need for targeted prevention strategies.

Stroke leads to significant mobility challenges, balance difficulties, and a diminished quality of life, making it the leading cause of walking and balance disabilities in older adults [8]. Approximately 75% of stroke survivors experience mobility limitations each year, with 40% requiring assistance for walking [9]. Among those who regain some independence, 60% face challenges with community ambulation [10]. The American Stroke Association notes that 87% of strokes are ischemic, causing symptoms such as paralysis, balance loss, and post-stroke cramping [11]. Many post-stroke individuals encounter substantial impairments in muscle strength, balance, and postural control due to decreased sensory feedback and weaker motor responses, which increase the risk of falls and functional limitations [12]. Balance issues often arise from reduced muscle power, coordination deficits, and impaired sensory integration. Motor deficits, including hemiparesis, affect about 80% of stroke survivors [13]. These balance problems stem from challenges in proprioception, trunk muscle strength, and coordination, which can restrict independence and lead to social isolation and depression [14]. A study by Rudberg et al. (2020) emphasized that balance and walking difficulties are major concerns for stroke patients, underscoring the necessity for effective rehabilitation strategies [15].

Rehabilitation programs focusing on strength and balance training are essential for improving functional outcomes. Evidence suggests that these interventions can enhance ambulation, mobility, and overall functional performance in stroke survivors [16, 17]. While supervised training under the guidance of a physical therapist has been shown to be effective, many stroke survivors and their caregivers prefer home-based exercises due to comfort, a sense of autonomy and lack of access to the training centers. Despite rapid changes, accessing consistent professional healthcare support remains crucial in Saudi Arabia. Patients face challenges due to limited resources, staffing shortages, and barriers that hinder recovery. Additionally, cultural perceptions and social stigma surrounding disability and gender segregation affects the willingness to seek help and follow rehabilitation programs, complicating the recovery efforts [18-20]. This study aims to investigate the comparative effects of supervised versus unsupervised strength and balance training on balance and functional performance in ambulatory stroke patients. The hypothesis is that compared to supervised training, unsupervised training under remote guidance can also achieve significant improvements in post-stroke patients. This research is crucial for developing effective rehabilitation protocols that cater to the needs of stroke survivors, particularly those who may have difficulty accessing consistent professional support. Understanding the impact of different training modalities on stroke recovery will help inform best practices in rehabilitation and ultimately enhance the quality of life for individuals living with the after effects of stroke.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 25 to 65 who had suffered a stroke between one and 24 months prior and were medically stable without complications were screened to be included in this study.

They should have scored 3 or lower on the Modified Ashworth Scale for muscle spasticity and reported lower limb pain levels of 5 or less on a 10-point visual analog scale.

They should have been able to tolerate 45 minutes of physical activity, including rest period, and walk independently for at least 40 meters, with or without assistive devices.

Exclusion Criteria:

* Those with a history of previous strokes, other neurological conditions, mobility issues, severe medical conditions, or significant visual field loss were excluded.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 12 weeks
  Berg Balance Scale assesses patient's balance through 14 tasks, scored from 0 to 4. A change of 4 points indicates a significant improvement in balance, particularly in elderly populations
Physiological cost index | 12 week
  Physiological Cost Index, evaluates the heart rate during rest and walking to assess the physiological cost of ambulation. It is calculated as the difference between walking heart rate and resting heart rate divided by the average walking speed.
6-minute walk distance test | 12 Week
  6-minute walk distance test, developed by the American Thoracic Society, measures aerobic capacity and endurance by recording the distance walked in six minutes, providing insights into functional capacity across various physiological systems
Short form-36 questionnaire | 12 Week
  36-Item Short Form Survey is a widely-used questionnaire assesses health-related quality of life across eight domains, including physical and emotional well-being. It is a validated tool for measuring overall health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Majmaah University, Al-Majmaah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to the principal investigator and furnished upon request.
Supporting Information: ICF
Time Frame: 4 week